CLINICAL TRIAL: NCT04062383
Title: Positive Psychology for Acute Coronary Syndrome Patients: A proof-of Concept Feasibility Trial
Brief Title: Positive Emotions After Acute Coronary Events at Northwestern University
Acronym: PEACE-NU
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: In-person recruitment deemed not feasible due to COVID
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Judith Moskowitz, Professor, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STU00208301
Record Dates: First submitted 2018-10-26; First posted 2019-08-20 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: ACS - Acute Coronary Syndrome
Keywords: ACS; Positive Psychology; Motivational Interviewing; Positive emotions
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Psychology, Positive; Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Positive Psychology + Motivational Interviewing (Experimental): Participants will complete weekly positive psychology exercises and will systematically set goals related to physical activity. Study trainers will review the positive psychology exercises on the phone each week and will use motivational interviewing techniques to facilitate goal setting.
  Interventions: Behavioral: Positive Psychology + Motivational Interviewing

INTERVENTIONS:
Behavioral: Positive Psychology + Motivational Interviewing — For the positive psychology portion of the intervention, the study trainer will (a) review the week's positive psychology exercise, (b) discuss the rationale of the next week's positive psychology exercise through a guided review of the positive psychology manual, and (c) assign the next week's positive psychology exercise. For the motivational interviewing portion, participants will (a) review their physical activity goal from the prior week, (b) discuss techniques for improving physical activity, and (c) set a physical activity goal for the next week. Study trainers will use motivational interviewing techniques to facilitate goal setting.

SUMMARY:
This study is a single-arm, 12-week trial to test the feasibility of a PP-MI intervention for patients recently admitted following ACS. PP-MI is a novel positive psychology-based health behavior intervention that is adapted for patients hospitalized for ACS. The intervention aims to cultivate positive emotions in this vulnerable population that could provide broad and significant health benefits, and may have distinct-and more powerful-effects than simply attempting to dampen negative emotions.

The primary aim is to assess whether the intervention exercises are feasible and linked with immediate boosts in positive affect upon completion. The secondary goal is to provide the research team with greater experience recruiting inpatients with an ACS, successfully completing intervention sessions, and administering psychological and medical assessments by phone.

DETAILED DESCRIPTION:
The initial study visit will occur in-person two weeks after discharge from the hospital. Participants will meet with a member of the study staff (the study "trainer") and complete self-report questionnaires assessing health behavior adherence and mental and physical health. Then, a study interventionist will provide a treatment manual for the positive psychology + motivational interviewing intervention, review the rationale for the initial exercise, and assign the first exercise. If the participant is in the positive psychology + motivational interviewing condition, the trainer will explain the rationale for both the positive psychology and goal-setting and motivational interviewing portions of the program, and will be assigned the first exercise. Participants will then be given an accelerometer, which they will be asked to wear for 7 days to ensure that they are comfortable with the device and that useable data can be obtained from the participant. Participants will then complete twelve 30-minute weekly phone sessions with a study trainer. The phone sessions primarily will include a review of the prior week's session content and a discussion of the rationale and assignment of the next week's exercise/assignment. Upon the completion of these calls, a blinded member of the study staff will call participants to administer self-report outcome measures. Participants will also be asked to wear an accelerometer at the follow-up timepoint as an objective measure of physical activity, which they will return by mail to the study staff.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients must meet at least two of three World Health Organization criteria for an acute MI: typical chest pain, elevated cardiac enzymes, and electrocardiographic changes consistent with MI. For UA, participants must have new-onset angina within 2 months, exacerbation of previous angina with rest or with minimal exercise, or angina within 2 weeks of MI.
* Suboptimal adherence to health behaviors: eligible patients must meet a total item score of <15 (suboptimal) based on three Medical Outcomes Study-Specific Adherence Scale (MOS SAS) items OR a total item score of 15 and a physical activity item score of <5.

Exclusion Criteria:

* Cognitive deficits, assessed via a 6-item cognitive screen,33 used to assess appropriate participation of medically ill patients in research studies and defined by a score of < 4.
* Medical conditions precluding interviews or likely to lead to death within 6 months, determined in consultation with the primary treatment team and Dr. James Flaherty.
* Individuals who have undergone coronary artery bypass surgery, or any open heart surgery, in the past 1 year.
* Inability to perform moderate to vigorous physical activity, as defined by an inability to walk without aid of an assistive device such as a walker or cane, OR inability to walk at a steady pace for at least 5 minutes without stopping.
* Inability to communicate in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
Number of intervention sessions completed by participants | 12 weeks
  Measured by number of intervention sessions completed by participants

SECONDARY OUTCOMES:
Change in physical activity | Baseline, 12 week
  As measured by accelerometer
Change in medication adherence | Baseline, 12 week
  Measured by SRMA, a two-item self-report medication adherence scale measuring percentage of time patients report taking their heart medications in the past one and two weeks.
Change in dietary adherence | Baseline, 12 week
  Measured by the MEDFICTS scale, a National Cholesterol Education Program-developed scale inquiring about saturated fat.
Change in positive affect | Baseline, 12 week
  Measured by the Positive and Negative Affect Schedule (PANAS)
Change in trait optimism | Baseline, 12 week
  Measured by the Life Orientation Test-Revised (LOT-R)
Change in state optimism | Baseline, 12 week
  Measured by the State Optimism Scale developed by Dr. Jeff Huffman
Change in anxiety | Baseline, 12 week
  Measured by the anxiety subscale of the Hospital Anxiety and Depression Scale (HADS-A)
Change in depression | Baseline, 12 week
  Measured by the depression subscale of the Hospital Anxiety and Depression Scale (HADS-D)
Change in physical function | Baseline, 12 week
  Measured by the Duke Activity Status Index (DASI)
Change in health-related quality of life | Baseline, 12 week
  Measured by the Short Form 12 (SF-12)
Change in adherence to health behaviors | Baseline, 12 week
  Measured by the three items from the Medical Outcomes Study-Specific Adherence Scale (MOS SAS)
Change in cardiac symptoms | Baseline, 12 week
  Measured by a checklist taken from the Women and Ischemia Syndrome Evaluation Study
Change in physical activity | Baseline, 12 week
  Measured by the self-report International Physical Activity Questionnaire (IPAQ)
Change in perceived stress | Baseline, 12 week
  Measured by the perceived stress scale (PSS-4) measure

CONTACTS AND LOCATIONS:
Overall Officials: Judith Moskowitz, PhD, MPH, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fredrickson BL. The role of positive emotions in positive psychology. The broaden-and-build theory of positive emotions. Am Psychol. 2001 Mar;56(3):218-26. doi: 10.1037//0003-066x.56.3.218. PMID 11315248
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Colberg SR, Sigal RJ, Fernhall B, Regensteiner JG, Blissmer BJ, Rubin RR, Chasan-Taber L, Albright AL, Braun B; American College of Sports Medicine; American Diabetes Association. Exercise and type 2 diabetes: the American College of Sports Medicine and the American Diabetes Association: joint position statement. Diabetes Care. 2010 Dec;33(12):e147-67. doi: 10.2337/dc10-9990. PMID 21115758
- [Background] Lee PH, Macfarlane DJ, Lam TH, Stewart SM. Validity of the International Physical Activity Questionnaire Short Form (IPAQ-SF): a systematic review. Int J Behav Nutr Phys Act. 2011 Oct 21;8:115. doi: 10.1186/1479-5868-8-115. PMID 22018588
- [Background] Lu M, Safren SA, Skolnik PR, Rogers WH, Coady W, Hardy H, Wilson IB. Optimal recall period and response task for self-reported HIV medication adherence. AIDS Behav. 2008 Jan;12(1):86-94. doi: 10.1007/s10461-007-9261-4. Epub 2007 Jun 19. PMID 17577653
- [Background] National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults (Adult Treatment Panel III). Third Report of the National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults (Adult Treatment Panel III) final report. Circulation. 2002 Dec 17;106(25):3143-421. No abstract available. PMID 12485966
- [Background] Bush K, Kivlahan DR, McDonell MB, Fihn SD, Bradley KA. The AUDIT alcohol consumption questions (AUDIT-C): an effective brief screening test for problem drinking. Ambulatory Care Quality Improvement Project (ACQUIP). Alcohol Use Disorders Identification Test. Arch Intern Med. 1998 Sep 14;158(16):1789-95. doi: 10.1001/archinte.158.16.1789. PMID 9738608
- [Background] Scheier MF, Carver CS, Bridges MW. Distinguishing optimism from neuroticism (and trait anxiety, self-mastery, and self-esteem): a reevaluation of the Life Orientation Test. J Pers Soc Psychol. 1994 Dec;67(6):1063-78. doi: 10.1037//0022-3514.67.6.1063. PMID 7815302
- [Background] Shifren K, Hooker K. Stability and change in optimism: a study among spouse caregivers. Exp Aging Res. 1995 Jan-Mar;21(1):59-76. doi: 10.1080/03610739508254268. PMID 7744171
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Hlatky MA, Boineau RE, Higginbotham MB, Lee KL, Mark DB, Califf RM, Cobb FR, Pryor DB. A brief self-administered questionnaire to determine functional capacity (the Duke Activity Status Index). Am J Cardiol. 1989 Sep 15;64(10):651-4. doi: 10.1016/0002-9149(89)90496-7. PMID 2782256
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] Krantz DS, Olson MB, Francis JL, Phankao C, Bairey Merz CN, Sopko G, Vido DA, Shaw LJ, Sheps DS, Pepine CJ, Matthews KA. Anger, hostility, and cardiac symptoms in women with suspected coronary artery disease: the Women's Ischemia Syndrome Evaluation (WISE) Study. J Womens Health (Larchmt). 2006 Dec;15(10):1214-23. doi: 10.1089/jwh.2006.15.1214. PMID 17199462